CLINICAL TRIAL: NCT05563701
Title: Evaluation of the LVivo Image Quality Scoring (IQS)
Status: Completed | Type: Observational
Sponsor: DiA Imaging Analysis Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CR2P0021
Record Dates: First submitted 2022-09-22; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Heart Diseases; Arrhythmia, Cardiac; Angina Pectoris; Unstable Angina; Lung Diseases; Congestive Heart Failure; Shock
Keywords: Echocardiography (Echo); Image Quality Scoring (IQS); Ultrasound (US); Point of Care (POC); 4CH (Four (4) Chamber of the heart view); LV (Left Ventricle); ER (Emergency Room); ICU (Intensive Care Unit); EF (Ejection Fraction)
MeSH Terms: conditions — Heart Diseases; Arrhythmias, Cardiac; Angina Pectoris; Angina, Unstable; Lung Diseases; Heart Failure; Shock; Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study includes two parts:

Part 1:

* 100 examinations of patient referred for echo evaluation, containing clips that were acquired from the 4CH apical view were collected retrospectively. Each study includes 10 clips that represent typical user scanning errors
* Offline evaluation of the system (by batch processing) shall be performed by comparing the system output to preliminary quality tagging by experienced sonographers

Part 2:

* Live scans of apical 4CH clips of patients with indication for POCUS examination will be performed by POC physicians
* LVivo IQS shall be used (on Lumify) during the scan for patients that meet inclusion criteria until 50 exams will be collected. 3 sec of each scan shall be saved, and Image quality score (IQS) shall be documented
* Saved scans shall be reviewed by an expert physician to determine whether they are clinically interpretable

DETAILED DESCRIPTION:
Part 1 Total of 424 examination were collected from two medical centers. Participants that were referred to routine echo examinations and signed an informed consent were enrolled to the study. The image acquisition was done using ultrasound devices available in the medical centers. In addition Lumify ultrasound device was supplied by the sponsor.

Each examination contained 10 clips, each representing a different scanning scenario where the image acquisition contained transitions between common user "acquisition error" to correctly acquired images.

The examinations in DICOM format and echo reports were collected after anonymization, the patient details were documented in a study log that was stored in the medical center.

The collected clips were tagged for image quality by experienced sonographers. The distribution of the collected data according to ultrasound devices, age, gender and LV function was analyzed.

The data was randomly split into training and clinical validation sets, such that the proportion of data according to data distribution was maintained and the data set for the clinical evaluation will contain 100 patient examinations.

The LVivo IQS algorithm will be applied to the clinical validation set automatically by batch processing. The image quality score provided by the LVivo IQS will be compared to the image quality tagging by the sonographers

Part 2 The trial is designed as a prospective multicenter study, enrolling 50 patients at two medical centers. In each medical center Lumify ultrasound devices on which the LVivo IQS demo software will be installed will be provided for image acquisition. The image acquisition will be done by POC medical doctors, at different stages of their internship, that received POCUS training during their medical studies and are using ultrasound devices in accordance with their routine workflow. The scans will be done in different POC units including ER, ICU and internal departments.

ELIGIBILITY:
Inclusion Criteria:

Part 1 Study:

1. Age ≥18
2. Referred to routine Echo examination

Part 2 Study:

1. Age ≥18
2. Indication for POCUS

Exclusion Criteria:

Part 1 Study:

1. Subjects who fail to meet any inclusion criteria

Part 2 Study:

1. Subjects who fail to meet any inclusion criteria
2. Image quality 1-2 according to ACEP June 2018 [11]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Part 1 Patients age ≥18 referred for echo evaluation
  Part 2 Patients age ≥18 with indication for POCUS examination
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Part 1: Overall agreement of 75% between image quality classification by LVivo IQS and the data tagging by experienced sonographers | Up to 24 weeks
Part 2: 80% of the Exams with image quality 3-5 by visual estimation, received at least "Medium" image quality by LVivo IQS | Up to 24 weeks
Part 2: 90% of these cases (when at least "Medium" image quality is indicated by LVivo IQS) are clinically interpretable | Up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka university medical center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johri AM, Galen B, Kirkpatrick JN, Lanspa M, Mulvagh S, Thamman R. ASE Statement on Point-of-Care Ultrasound during the 2019 Novel Coronavirus Pandemic. J Am Soc Echocardiogr. 2020 Jun;33(6):670-673. doi: 10.1016/j.echo.2020.04.017. Epub 2020 Apr 15. PMID 32503704
- [Background] Hashim A, Tahir MJ, Ullah I, Asghar MS, Siddiqi H, Yousaf Z. The utility of point of care ultrasonography (POCUS). Ann Med Surg (Lond). 2021 Nov 2;71:102982. doi: 10.1016/j.amsu.2021.102982. eCollection 2021 Nov. No abstract available. PMID 34840746
- [Background] Dall T. et al. The Complexities of Physician Supply and Demand: Projections From 2019 to 2034. Association Of American Medical Collage, 2021.
- [Background] Blanco P, Volpicelli G. Common pitfalls in point-of-care ultrasound: a practical guide for emergency and critical care physicians. Crit Ultrasound J. 2016 Dec;8(1):15. doi: 10.1186/s13089-016-0052-x. Epub 2016 Oct 26. PMID 27783380
- [Background] Smistad E, Ostvik A, Salte IM, Melichova D, Nguyen TM, Haugaa K, Brunvand H, Edvardsen T, Leclerc S, Bernard O, Grenne B, Lovstakken L. Real-Time Automatic Ejection Fraction and Foreshortening Detection Using Deep Learning. IEEE Trans Ultrason Ferroelectr Freq Control. 2020 Dec;67(12):2595-2604. doi: 10.1109/TUFFC.2020.2981037. Epub 2020 Nov 24. PMID 32175861
- [Background] Unlu S, Duchenne J, Mirea O, Pagourelias ED, Bezy S, Cvijic M, Beela AS, Thomas JD, Badano LP, Voigt JU; EACVI-ASE Industry Standardization Task Force. Impact of apical foreshortening on deformation measurements: a report from the EACVI-ASE Strain Standardization Task Force. Eur Heart J Cardiovasc Imaging. 2020 Mar 1;21(3):337-343. doi: 10.1093/ehjci/jez189. PMID 31361311
- [Background] Kumar V. There is No Substitute for Human Intelligence. Indian J Crit Care Med. 2021 May;25(5):486-488. doi: 10.5005/jp-journals-10071-23832. PMID 34177163
- [Background] Narang A, Bae R, Hong H, Thomas Y, Surette S, Cadieu C, Chaudhry A, Martin RP, McCarthy PM, Rubenson DS, Goldstein S, Little SH, Lang RM, Weissman NJ, Thomas JD. Utility of a Deep-Learning Algorithm to Guide Novices to Acquire Echocardiograms for Limited Diagnostic Use. JAMA Cardiol. 2021 Jun 1;6(6):624-632. doi: 10.1001/jamacardio.2021.0185. PMID 33599681
- [Background] Liu B.R et al. Emergency Ultrasound Standard Reporting Guidelines. ACEP, 2018. pp. 2-44.
- [Background] Dixon, W.J., Massey, F.J. Introduction to Statistical Analysis. 4th Edition McGraw-Hill, 1983. pp. 105-107
- [Background] Nagata Y, Kado Y, Onoue T, Otani K, Nakazono A, Otsuji Y, Takeuchi M. Impact of image quality on reliability of the measurements of left ventricular systolic function and global longitudinal strain in 2D echocardiography. Echo Res Pract. 2018 Mar;5(1):27-39. doi: 10.1530/ERP-17-0047. Epub 2018 Feb 5. PMID 29432198
- [Background] Russell FM, Herbert A, Ferre RM, Zakeri B, Echeverria V, Peterson D, Wallach P. Development and implementation of a point of care ultrasound curriculum at a multi-site institution. Ultrasound J. 2021 Feb 21;13(1):9. doi: 10.1186/s13089-021-00214-w. PMID 33615390
- [Background] Goldman, L. et al. Echocardiography. Elsevier, Inc, 2020. pp. 253-260
- See also: EchoNous official cite — https://echonous.com/en_us/
- See also: Ultrasight official site — https://www.ultrasight.com/